CLINICAL TRIAL: NCT03418467
Title: Evaluation of Risk Factors for Therapeutic Outcome in Patients with Tachycardiomyopathy
Brief Title: Risk Factors in Tachycardiomyopathy
Acronym: EMPATHY
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: EMPATHY-1
Record Dates: First submitted 2018-01-24; First posted 2018-02-01 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Atrial Fibrillation; Atrial Flutter; Ventricular Premature Complexes
Keywords: Tachycardiomyopathy; atrial fibrillation; EMID (enrichment of mitochondria at the intercalated discs); Biopsy; empathy
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter; Ventricular Premature Complexes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- tachycardiomyopathy: Sustained heart rate of over 100 bpm, exclusion of other causes of congestive heart failure including significant valvular disease and coronary artery stenosis over 50%, and partial or complete recovery of left ventricular function after restoration of sinus rhythm or rate control and characteristic histological findings.
- dilated cardiomyopathy: Patients with dilated cardiomyopathy according to the 2016 ESC (European Heart Association) Guidelines for the diagnosis and treatment of acute and chronic heart failure.

SUMMARY:
Decision between rate control and rhythm control can be a challenge in clinical practice. While there is some guiding evidence, we still lack a comprehensive insight into different subgroups of patients that will benefit from a rhythm control treatment.

EMPATHY is a prospective clinical study in patients presenting with heart failure and a tachyarrhythmic rhythm disturbance. Biomarkers, routinely obtained results from clinical examinations, and results from endomyocardial biopsies shall be evaluated to identify patients which have better outcome from a rhythm control strategy by ablation therapy or, if contraindicated by pharmacological rhythm control.

This study is designed to identifying risk factors and subgroups profiting from rhythm restoration and therefore improve current therapeutic approaches and the rate of recurrence-free survival.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed left ventricular ejection fraction ≤ 50%
* endomyocardial biopsy available
* tachycardic rhythm disturbance with a rhythm control strategy planned for tachycardic atrial fibrillation or flutter (≥100/min) or more than 10000 ventricular premature beats in 24 hours

Exclusion Criteria:

* age <18 years
* patient unable or unwilling to give informed consent
* coronary artery stenosis >50%
* relevant valvular disease
* simultaneous contraindications against amiodarone treatment and pulmonary vein isolation/ablation therapy
* present or suspected alcohol/drug dependency will result in exclusion from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting at the University Hospital Tübingen with decreased left ventricular ejection fraction.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-10-11 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
histological characteristics | 3 months
  Identification of histopathological criteria, which indicate better outcome after rhythm control. Recovery of left ventricular ejection fraction (assessed by echocardiography) will be measured.

SECONDARY OUTCOMES:
recurrence of rhythm disturbance | 3 months
  Evaluating the recurrence of the underlying rhythm disturbance (ECG, 7 day holter monitoring, implantable event recorder)
rehospitalization | 3 months
  Evaluating the rate of unplanned rehospitalization
all-cause mortality | 3 months
  Evaluating the all-cause mortality
NYHA class (New York Heart Association) | 3 months
  Evaluating the extend of heart failure symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Tübingen, Medizinische Klinik III (Kardiologie), Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No